CLINICAL TRIAL: NCT06387680
Title: The Effect of Peanut Ball Use on Labor Memory, Labor Satisfaction, Delivery Length, and Neonatal APGAR Score: A Randomized Controlled Trial
Brief Title: The Peanut Ball Use on Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Seyhan Çankaya, Assoc. Prof. Seyhan Çankaya, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/187
Record Dates: First submitted 2024-04-16; First posted 2024-04-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Birth Outcome, Adverse; Birth, First; Labor Long; Apgar; 4-7 at 1 Minute
Keywords: Birth memory and recall; Birth satisfaction; Labor length; APGAR score; Peanut ball
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut Ball Group (Experimental): When the cervical dilation reached 4 cm, the peanut ball was first applied to the pregnant women in the side-lying position (right side/left side) for 20 minutes, and then the pregnant women were allowed to rest for 10 minutes. Second, the semi-seated position was applied for 20 minutes and the pregnant women were allowed to rest for 10 minutes. Third, the supine position was applied for 20 minutes followed by 10 minutes of rest. Fourth, the hand-knee position was applied for 20 minutes and rested for 10 minutes. Finally, the squatting position was practiced for 20 minutes and then the pregnant women rested for 10 minutes. Each position was practiced with the peanut ball for 20 minutes and rested for 10 minutes. Each position was performed once during the procedure. A pregnant woman who wished to remain in a position longer was allowed an additional 10 minutes without interrupting the flow of the intervention and then rested for 10 minutes.
  Interventions: Other: The Effect of Peanut Ball Use on Labor Memory, Labor Satisfaction, Delivery Length, and Neonatal APGAR Score: A Randomized Controlled Trial
- Control Group (No Intervention): Control Group (CG) No intervention other than routine intrapartum midwifery care was provided to primiparous pregnant women in the control group. After admission to the hospital for delivery, the pregnant women in the control group were informed about the study, written informed consent was obtained, routine practices and care in the delivery room were performed (taking history, taking vital signs, demonstrating correct breathing techniques, ensuring freedom of movement), vaginal examination and cervical changes were recorded on the partograph, EFM (electronic fetal monitoring) was performed when the time came according to the doctor's order, fetal heart rate (FHR) was listened to every half hour and recorded on the partograph.

INTERVENTIONS:
Other: The Effect of Peanut Ball Use on Labor Memory, Labor Satisfaction, Delivery Length, and Neonatal APGAR Score: A Randomized Controlled Trial — The Effect of Peanut Ball Use on Labor Memory, Labor Satisfaction, Delivery Length, and Neonatal APGAR Score: A Randomized Controlled Trial
  Arms: Peanut Ball Group

SUMMARY:
The purpose of this study was to evaluate the effect of using peanut balls during labor on labor memory, labor satisfaction, labor length, and neonatal APGAR scores.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the effect of using peanut balls during labor on labor memory, labor satisfaction, labor length, and neonatal APGAR scores.

This randomized, controlled, single-blind trial was conducted in 156 primiparous pregnant women (peanut ball group n=78, control group n=78) who delivered between March 2024 and October 2024. Pregnant women in the peanut ball group were instructed to perform movements with the peanut ball after cervical dilation reached 4 cm. The control group received only standard intrapartum midwifery care. Data were collected by personal information form, labor and postpartum follow-up form (APGAR score, etc.), Birth Memory and Recall Scale 4 hours after delivery, and Birth Satisfaction Scales.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women were included if they had indications for vaginal delivery,

* Were primiparous,
* Had cervical dilation of 3 cm or more,
* Had term pregnancy (38 to 42 weeks of gestation),
* Had a single,
* Healthy,
* Vertex-positioned fetus,
* Had no complications that could cause dystocia during labor (contraction anomalies, birth object, dystocia related to the birth canal, dystocia related to the mother's psyche, dystocia related to the mother's psychology),
* Did not use analgesia and anesthesia during the first stage of labor,
* I did not have any physical disability to take the positions to be used in the study,
* Did not have any communication problems,
* Had language skills sufficient to speak and understand Turkish.

Exclusion Criteria:

* Pregnant women were excluded if they had abnormal changes in fetal heart rate during labor (fetal distress, etc.),
* Had an unexpected pregnancy or fetal complication,
* Had a high-risk pregnancy,
* Were taking magnesium sulfate,
* Had symptoms of intrauterine infection,
* Had previously attended antenatal classes,
* Or reported having been educated about birthing balls.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of sociodemographic of pregnant women. | 6 months
  Sociodemographic of pregnant women will be collected through surveys and compared and reported.
Comparison of obstetric characteristics of pregnant women | 6 months
  Obstetric of pregnant women will be collected through surveys and compared and reported.
Comparison of postpartum characteristics of pregnant women | 6 months
  Postpartum characteristics of pregnant women will be collected through surveys and compared and reported.
Comparison of duration of 1st and 2nd stage of labor by group | 6 months
  The 1st and 2nd stages of the birth of pregnant women will be followed by the midwife and notes will be taken in the survey.
Comparison of 1st and 5th minute APGAR scores of newborns by group | 6 months
  The 1st and 5th minute APGAR scores of newborns will be noted in the survey.
Comparison of the mean scores of the Pregnant Women's Birth Memory and Recall Questionnaire (BirthMARQ) and its subscales by groups | 6 months
  BirthMARQ scale will be applied to pregnant women. BirthMARQ ranges from 1 to 147 points (min-max), with higher scores indicating poor mood and more frequent involuntary recall.
Comparison of pregnant women's Birth Satisfaction Scale (BSS) mean scores by groups | 6 months
  BSS scale will be applied to pregnant women.BSS is 0-40 points (min-max), and as the score increases, the level of birth satisfaction increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Cankaya S, Alan Dikmen H, Atas A. The effect of peanut ball use on labor memory, labor satisfaction, delivery length, and neonatal APGAR score: a randomized controlled trial. Postgrad Med. 2025 Jun;137(5):368-378. doi: 10.1080/00325481.2025.2510198. Epub 2025 May 26. PMID 40396494